CLINICAL TRIAL: NCT01478516
Title: Autologous Intravitreal Plasmin and Fibrinolytic System of Vitreous in Patient With Macular Edema
Brief Title: Autologous Plasmin and Fibrinolytic System in Diabetic Retinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Collaborators: Hallym University (Other)
Responsible Party: Principal Investigator, Jiwon Lim, MD PhD, Hallym University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-72
Record Dates: First submitted 2011-11-17; First posted 2011-11-23 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Macular Edema
Keywords: autologous plasmin; macular edema; vitreous
MeSH Terms: conditions — Macular Edema | interventions — Intravitreal Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Plasmin (Experimental): eyes with macular edema
  Interventions: Procedure: Intravitreal injection

INTERVENTIONS:
Procedure: Intravitreal injection — autologous plasmin was prepared in the operation department. Samples (3.5 mL) of autologous whole blood, collected by sterile vacuum blood collection tubes, were obtained from a peripheral vein. The blood was centrifuged at 4,000 rounds per minute for 15 minutes to obtain complete sedimentation of the cells; 1.5 mL of the plasma was aspirated and transferred under sterile conditions in a vial of urokinase(10,000 IU) that had been incubated for 15 minutes at 37°C. By gently moving the vial for 5 minutes, the solution was incubated for 15 minutes at 37°C; 0.2 mL of the obtained solution was used for intravitreal injection.

SUMMARY:
The purpose of this study is to evaluate in a prospective study the efficacy of intravitreal autologous plasmin enzyme in macular edema and to analyze the fibrinolytic system in vitreous body.

DETAILED DESCRIPTION:
Autologous plasmin enzyme has been used to liquefy the gel structure of the vitreous body and to decrease the adherence of the posterior vitreous cortex to the inner limiting membrane in clinical studies. The investigators performed intravitreal autologous plasmin enzyme for macular edema. in addition, the investigators collected vitreous body in macular edema and analyzed fibrinolytic system.

ELIGIBILITY:
Inclusion Criteria:

* eyes with macular edema
* those who showed poor outcomes in visual acuity or macular thickness after grid laser,triamcinolone,or bevacizumab therapy or a combination of these treatments.

Exclusion Criteria:

* uncontrolled blood pressure (systolic and diastolic blood pressure greater than 150 and 90 mm Hg, respectively)
* renal insufficiency
* intraocular surgery or any intravitreal treatment during the previous 3 months
* history of ocular hypertension and/or glaucoma

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Central macular thickness after intravitreal autologous plasmin injection | 1 month after intervention
  Central macular thickness measured by optocal coherence tompgraphy
Visual acuity after intravitreal autologous plasmin | 1 Month after intervention
  logMAR visual acuity

SECONDARY OUTCOMES:
fibrinolytic system | baseline
  plasminogen, tissue plasminogen activetor, anti-pasminogen receptor, antithrombin

CONTACTS AND LOCATIONS:
Overall Officials: Jiwon Lim, MDPhD, Principal Investigator — Chuncheon Sacred Heart Hospital
Locations (1):
- Ji Won Lim, Chuncheon, Gangwon-do, South Korea